CLINICAL TRIAL: NCT02232087
Title: Phase I Single Blind, Randomised, Cross-over Pharmacodynamic Dose Response Study in Healthy Volunteers of Two Pressurized Metered Dose Inhalers (pMDIs) That Deliver Salmeterol and Fluticasone Propionate
Brief Title: Single Blind Cross-over Dose Response Study in Subjects of Two Inhalers of Salmeterol and Fluticasone Propionate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kindeva Drug Delivery (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: DDSD-1030-SAFL
Record Dates: First submitted 2014-09-02; First posted 2014-09-04 (Estimated); Results first posted 2020-11-02 (Actual); Last update posted 2022-06-15 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: long-acting beta agonist (LABA); corticosteroid; pMDI; inhaler
MeSH Terms: interventions — Salmeterol Xinafoate; Fluticasone

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- test product A (Experimental): salmeterol and fluticasone propionate, 2 puffs
  Interventions: Drug: Salmeterol; Drug: fluticasone propionate
- reference product D (Active Comparator): salmeterol and fluticasone propionate, 2 puffs
  Interventions: Drug: Salmeterol; Drug: fluticasone propionate
- test product B (Experimental): salmeterol and fluticasone propionate, 6 puffs
  Interventions: Drug: Salmeterol; Drug: fluticasone propionate
- reference product E (Active Comparator): salmeterol and fluticasone propionate, 6 puffs
  Interventions: Drug: Salmeterol; Drug: fluticasone propionate
- test product C (Experimental): salmeterol and fluticasone propionate, 12 puffs
  Interventions: Drug: Salmeterol; Drug: fluticasone propionate
- reference product F (Active Comparator): salmeterol and fluticasone propionate, 12 puffs
  Interventions: Drug: Salmeterol; Drug: fluticasone propionate

INTERVENTIONS:
Drug: Salmeterol — A, D 2 puffs; B, E 6 puffs; C, F 12 puffs
  Other Names: Sirdupla; Seretide Evohaler
Drug: fluticasone propionate — A, D 2 puffs; B, E 6 puffs; C, F 12 puffs
  Other Names: Sirdupla; Seretide Evohaler

SUMMARY:
The purpose of this study is to test the body's response to several doses of two different inhalation products in healthy volunteers.

DETAILED DESCRIPTION:
Healthy subjects will be enrolled and will receive 2, 6, and 12 inhalations from both the test and reference pMDI products according to a six-period cross-over design. Electrocardiograms (ECGs) and plasma potassium and glucose levels will be measured pre-dose and over 6 hours post-dose.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Volunteer
* Willing and able to give informed consent
* Willing to withhold all alcoholic beverages for 48 hours and all xanthine- containing foods and beverages for 24 hours prior to reporting to clinic
* Male and female subjects aged 18 to 55 years (inclusive)
* Subjects must agree to use an adequate method of contraception from admission through 12 weeks after last administration

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities or disease or chronic respiratory disorders
* Any presence or history of a clinically significant allergy including any adverse reaction to study drug
* History of drug or alcohol abuse within the past 2 years
* Smoked tobacco within the past 6 months or have a history of more than 10- pack years (number of packs smoked per day x number of years smoked)
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Have received any prescription medication within 4 weeks or investigational medication within 12 weeks of study (exception: contraceptives are permitted)
* Have received any non-prescription medication within 14 days prior to dosing (exception: paracetamol use within 2 days)
* Upper respiratory tract infection (excluding otitis media) within 14 days of the first study day, or lower respiratory tract infection within the last 3 months
* If female, nursing, lactating or pregnant
* Regular alcohol consumption in males >21 units per week and females >14 units per week (1 unit = ½ pint beer, 25 mL of 40% spirit or a 125 mL glass of wine)
* Surgery scheduled during the study or within 3 weeks after last dose
* History of familial long QT syndrome or history of sudden death in family members aged < 30 years

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2014-07; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pui Leung, MD, Principal Investigator — Quotient Clinical Ltd
Locations (1):
- Quotient Clinical Ltd, Ruddington, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Harrison LI, Sessions V, Wiggenhorn CJ, Chalmers D, Leung P, Efthimiou J. Comparison of systemic pharmacodynamic effects of two combination pressurized metered dose inhalers that deliver salmeterol and fluticasone propionate. Br J Clin Pharmacol. 2017 Nov;83(11):2377-2385. doi: 10.1111/bcp.13349. Epub 2017 Aug 1. PMID 28626983

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began 07 July 2014
Groups:
- Sequence 1 (A, F, B, E, C, D); Sequence 2 (B, A, C, F, D, E); Sequence 3 (C, B, D, A, E, F); Sequence 4 (D, C, E, B, F, A); Sequence 5 (E, D, F, C, A, B); Sequence 6 (F, E, A, D, B, C ): salmeterol and fluticasone propionate per inhalation
  A = 2 inhalations (test product), B = 6 inhalations (test product), C = 12 inhalations (test product), D = 2 inhalations (reference product), E = 6 inhalations (reference product) and F = 12 inhalations (reference product)
Period: Overall Study
Arm/Group | Sequence 1 (A, F, B, E, C, D) | Sequence 2 (B, A, C, F, D, E) | Sequence 3 (C, B, D, A, E, F) | Sequence 4 (D, C, E, B, F, A) | Sequence 5 (E, D, F, C, A, B) | Sequence 6 (F, E, A, D, B, C )
Started | 9 | 10 | 8 | 8 | 8 | 9
Completed | 7 | 8 | 8 | 7 | 7 | 6
Not Completed | 2 | 2 | 0 | 1 | 1 | 3
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 0 | 1
Not completed — poor inhalation technique | 0 | 1 | 0 | 0 | 0 | 2
Not completed — protocol stop criteria | 0 | 1 | 0 | 1 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: all subjects who received at least one test and one reference product for same dose
Groups:
- All Subjects: salmeterol and fluticasone propionate
Arm/Group | All Subjects
Number analyzed (Participants) | 52
Age, Continuous [Mean (Standard Deviation); unit: years] — age range of 18 to 55 years inclusive
  years | 33.5 (10.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23
  Male | 29
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 46
  More than one race | 0
  Unknown or Not Reported | 4
Region of Enrollment [Number; unit: participants]
  United Kingdom | 52
BMI [Mean (Standard Deviation); unit: kg/m2] | 23.6 (1.8)
forced expiratory volume at one second [Mean (Standard Deviation); unit: % predicted normal] — forced expiratory volume at one second > 85% predicted
  % predicted normal | 101.19 (10.74)

OUTCOME MEASURES:

1. Primary Outcome: Relative Potency Max Heart Rate
Description: Selection of steepest part of dose response curve for Relative Potency: 6 and 12 inhalation dose pairs. Slope of B and C line compared with slope of E and F to obtain relative potency value. Two inhalation dose not utilized as not on steepest part of curve.
Time Frame: Baseline, up to 6 hrs
Population: relative potency calculated for dose pairs B (6 inhalations) and C (12 inhalations), compared with E (6 inhalations) and F (12 inhalations)
Measure: Number (90% Confidence Interval); unit: unitless
Groups:
- Test B and C vs Reference E and F: salmeterol and fluticasone propionate
  Salmeterol: B, E 6 puffs; C, F 12 puffs
  fluticasone propionate: B, E 6 puffs; C, F 12 puffs
Arm/Group | Test B and C vs Reference E and F
Number analyzed (Participants) | 42
unitless | 0.8619 [0.7209 to 1.00]
Statistical Analysis 1: Comparison: Test B and C vs Reference E and F; The measurement of relative potency was conducted for the pair of doses which met the above criteria and lay on the steepest linear portion of the dose response curve. The log estimate of relative potency was obtained as the ratio of the estimated treatment effect as measured by the difference in the intercepts of the parallel lines divided by the estimate of the common slope for log dose; Test type: Equivalence — The potency of the test and reference product was considered equivalent if the 90% CI for the estimate of relative potency was completely contained within the limits of 0.67 to 1.50; p > 0.10, ANOVA — test for parallelism of dose response lines; Odds Ratio, log = 1.00, 90% CI 2-sided [0.67 to 1.50] — Test is the numerator

2. Primary Outcome: Relative Potency QTcB Interval
Description: Selection of steepest part of dose response curve for Relative Potency: 2 and 6 inhalation dose pairs. Slope of A and B line compared with slope of D and E to obtain relative potency value. Twelve inhalation dose not utilized as not on steepest part of curve.
Time Frame: Baseline up to 6 hrs
Population: relative potency calculated for dose pairs A (2 inhalations) and B (6 inhalations), compared with D (2 inhalations) and E (6 inhalations)
Measure: Number (90% Confidence Interval); unit: unitless
Groups:
- Test A and B vs Reference D and E: salmeterol and fluticasone propionate
  Salmeterol: A, D 2 puffs; B, E 6 puffs
  fluticasone propionate: A, D 2 puffs; B, E 6 puffs
Arm/Group | Test A and B vs Reference D and E
Number analyzed (Participants) | 42
unitless | 1.0760 [0.8206 to 1.4238]
Statistical Analysis 1: Comparison: Test A and B vs Reference D and E; [analysis description as in outcome 1, analysis 1]; Test type: Equivalence — [test comment as in outcome 1, analysis 1]; p > 0.10, ANOVA — test for parallelism of dose response lines; Odds Ratio, log = 1.00, 90% CI 2-sided [0.67 to 1.50] — Test is the numerator

3. Secondary Outcome: Max Heart Rate
Description: max heart rate at the 2, 6, or 12 inhalations dose, assessed at multiple times over 6 hours
Time Frame: Baseline through 6 hours
Population: subjects who received the test and the reference product at the 2, 6, or 12 inhalations dose
Measure: Mean (Standard Deviation); unit: bpm
Groups:
- Test Product A; Reference Product D: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 2 inhalations
  fluticasone propionate: 2 inhalations
- Test Product B; Reference Product E: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 6 inhalations
  fluticasone propionate: 6 inhalations
- Test Product C: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 12 inhalations
  fluticasone propionate: 12 inhalations
- Reference Product F: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate):12 inhalations
  fluticasone propionate: 12 inhalations
Arm/Group | Test Product A | Reference Product D | Test Product B | Reference Product E | Test Product C | Reference Product F
Number analyzed (Participants) | 43 | 43 | 45 | 45 | 44 | 46
bpm | 65.1 (10.9) | 65.5 (10.1) | 68.9 (11.0) | 69.9 (12.2) | 75.3 (13.3) | 76.8 (14.8)
Statistical Analysis 1: Comparison: Test Product A vs Reference Product D; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.55, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-2.5 to 1.4] — Comparability confirmed if confidence interval includes zero
Statistical Analysis 2: Comparison: Test Product B vs Reference Product E; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.53, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 1.0, 95% CI 2-sided [-2.5 to 1.3] — Comparability confirmed if confidence interval includes zero
Statistical Analysis 3: Comparison: Test Product C vs Reference Product F; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.011, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 1.00, 95% CI 2-sided [-2.5 to 1.3] — Comparability confirmed if confidence interval includes zero

4. Secondary Outcome: Plasma Potassium Level
Description: maximum plasma levels of potassium at 2, 6 or 12 inhalations dose inhalations dose, assessed a multiple times over 6 hours.
Time Frame: baseline through 6 hours
Population: subjects who received both the test and reference products at the 2, 6, or 12 inhalations dose
Measure: Mean (Standard Deviation); unit: mmol/L
Groups:
- Test Product A: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 2, 6, and 12 inhalations
  fluticasone propionate: 2 inhalations
- Reference Product F: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 12 inhalations
  fluticasone propionate: 12 inhalations
Arm/Group | Test Product A | Reference Product D | Test Product B | Reference Product E | Test Product C | Reference Product F
Number analyzed (Participants) | 43 | 43 | 45 | 45 | 44 | 46
mmol/L | 3.82 (0.19) | 3.78 (0.16) | 3.76 (0.20) | 3.75 (0.19) | 3.63 (0.24) | 3.61 (0.26)
Statistical Analysis 1: Comparison: Test Product A vs Reference Product D; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.26, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.03 to 0.10] — Comparability confirmed if confidence interval includes zero
Statistical Analysis 2: Comparison: Test Product B vs Reference Product E; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.93, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.06 to 0.06] — Comparability confirmed if confidence interval includes zero
Statistical Analysis 3: Comparison: Test Product C vs Reference Product F; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.48, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.04 to 0.08] — Comparability confirmed if confidence interval includes zero

5. Secondary Outcome: Max Plasma Glucose Level
Description: maximum levels of glucose at the 2, 6 or 12 inhalations dose, assessed at multiple times over 6 hours.
Time Frame: baseline through 6 hours
Population: subjects who received both the test and reference products at the two inhalations dose
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Test Product A | Reference Product D | Test Product B | Reference Product E | Test Product C | Reference Product F
Number analyzed (Participants) | 43 | 43 | 45 | 45 | 44 | 46
mmol/L | 5.31 (0.49) | 5.31 (0.40) | 5.53 (0.65) | 5.62 (0.54) | 5.88 (0.66) | 5.98 (0.65)
Statistical Analysis 1: Comparison: Test Product A vs Reference Product D; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.93, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0 — Comparability confirmed if confidence interval includes zero
Statistical Analysis 2: Comparison: Test Product B vs Reference Product E; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.42, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.224 to 0.093] — Comparability confirmed if confidence interval includes zero
Statistical Analysis 3: Comparison: Test Product C vs Reference Product F; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.078, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-0.302 to 0.016] — Comparability confirmed if confidence interval includes zero

6. Secondary Outcome: Max QTcB
Description: For each dose, the 95% CIs for the mean difference for the test product versus the reference product were calculated.
Time Frame: Baseline through 6 hours
Population: all subjects who received the test and the reference product at the two inhalations dose
Measure: Mean (Standard Deviation); unit: ms
Groups:
- Test Product D; Reference Product F: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 12 inhalations
  fluticasone propionate: 12 inhalations
Arm/Group | Test Product A | Reference Product D | Test Product B | Reference Product E | Test Product D | Reference Product F
Number analyzed (Participants) | 43 | 43 | 45 | 45 | 44 | 46
ms | 422.3 (22.4) | 422.1 (23.7) | 430.0 (23.1) | 430.2 (21.4) | 441.0 (20.5) | 444.0 (26.7)
Statistical Analysis 1: Comparison: Test Product A vs Reference Product D; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.71, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-3.9 to 5.7] — Comparability confirmed if confidence interval includes zero
Statistical Analysis 2: Comparison: Test Product B vs Reference Product E; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 1.00, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = 0, 95% CI 2-sided [-4.7 to 4.7] — Comparability confirmed if confidence interval includes zero
Statistical Analysis 3: Comparison: Test Product D vs Reference Product F; For each dose, the 95% CIs for the mean differences for the test product versus the reference product were calculated; Test type: Equivalence — Comparability confirmed if confidence interval includes zero; p = 0.016, ANOVA — Comparability demonstrated for p>0.05; Mean Difference (Final Values) = -2, 95% CI 2-sided [-10.6 to -1.1] — Comparability confirmed if confidence interval includes zero

ADVERSE EVENTS:
Time Frame: Adverse events were collected for up to 2 months for each subject. The duration of the clinical phase of the study was 4 months.
Description: All subjects who received a dose of at least one product
Groups:
- Reference Product D: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 6 inhalations
  fluticasone propionate: 6 inhalations
- Reference Product E: salmeterol and fluticasone propionate
  salmeterol (as salmeterol xinafoate): 12 inhalations
  fluticasone propionate: 12 inhalations
- Referencet Product F: salmeterol and fluticasone propionate
Arm/Group | Test Product A | Test Product B | Test Product C | Reference Product D | Reference Product E | Referencet Product F
All-Cause Mortality (participants affected / at risk) | 4/49 | 5/48 | 11/47 | 5/47 | 4/48 | 8/50
Serious Adverse Events (participants affected / at risk) | 0/49 | 0/48 | 0/47 | 0/47 | 0/48 | 0/50
Other Adverse Events (participants affected / at risk) | 4/49 | 5/48 | 11/47 | 5/47 | 4/48 | 8/50
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Test Product A (N=49) | Test Product B (N=48) | Test Product C (N=47) | Reference Product D (N=47) | Reference Product E (N=48) | Referencet Product F (N=50)
headache (Nervous system disorders) | 2 | 2 | 4 | 3 | 4 | 4
Asthenia (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mouth Ulceration (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 1 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 1
Feeling Hot (General disorders) | 0 | 0 | 0 | 0 | 1 | 2
Feeling Cold (General disorders) | 0 | 0 | 1 | 0 | 0 | 0
ECG QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 1
Prolongation (Investigations) | 0 | 0 | 1 | 0 | 0 | 0
Heart Rate increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 2
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1 | 0
tremor (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 4 | 0 | 0 | 0
Nervousness (Psychiatric disorders) | 0 | 0 | 1 | 0 | 1 | 3
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Rhinorrtoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 2
URTI (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Paraesthesia Oral (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0

LIMITATIONS AND CAVEATS:
There are no limitations or caveats.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor reserves the right to the first publication of the results. Following the first publication, or if the sponsor confirms in writing no interest in publishing the results, Quotient Clinical Ltd or the Principal Investigator may proceed to publish results from the study, giving the sponsor 60 days to review the manuscript.